# **Cover Page**

**Document:** Informed Consent Form

Official Study Title: Achieving Nutritional Adequacy Of Vitamin E With An

Egg/Plant-Based Food Pairing

ClinicalTrials.gov ID: NCT04287816

## **Document Date:**

• Informed Consent Form Study-1: 12/07/2020

• Informed Consent Form Study-2: 12/07/2020

• Informed Consent Form Study-3: 07/28/2022

IRB Approval date:

Version: Ver 2 (Dec 7,

2020)

# The Ohio State University Consent to Participate in Research

Study Title: Achieving Nutritional Adequacy Of Vitamins E and K With An

Egg/Plant-Based Food Pairing – Study 1

**Principal Investigator:** Richard S. Bruno

**Sponsor:** Egg Nutrition Center / American Egg Board

- This is a consent form for research participation. It contains important information about this study and what to expect if you decide to participate. Please consider the information carefully. Feel free to discuss the study with your friends and family and to ask questions before making your decision whether or not to participate.
- Your participation is voluntary. You may refuse to participate in this study. If you decide to take part in the study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your usual benefits. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.
- You may or may not benefit as a result of participating in this study. Also, as explained below, your participation may result in unintended or harmful effects for you that may be minor or may be serious depending on the nature of the research.
- You will be provided with any new information that develops during the study that may affect your decision whether or not to continue to participate. If you decide to participate, you will be asked to sign this form and will receive a copy of the form. You are being asked to consider participating in this study for the reasons explained below.

#### **Key Information About This Study**

The following is a short summary to help you decide whether or not to be a part of this study. More detailed information is listed later in this form.

The purpose of this research is to understand how the absorption of vitamin E and vitamin K found in vegetables like spinach can be improved when eaten along with other foods like eggs that contain fat. If you choose to participate in this study, your involvement would span approximately 12 weeks. During this period, there will be 6 nutrient absorption trials. Each trial would last 72 hours and a trained individual would be collecting blood samples periodically from your arm (11 in total). However, you will be free to come and go from our study center during each trial. The primary risk in this study relates to the small initial pain, bruising, or lightheadedness you may experience during blood collection. There are no costs to you to participate in this research and benefits to you include receiving some of your blood testing results like glucose along with your blood pressure and body mass measurements.

IRB Approval date:


2020)

## 1. Why is this study being done?

Vitamin E and vitamin K are two important nutrients for human health. However, the majority of Americans eat diets that are lacking in these nutrients. In addition, when we eat vegetables containing these high levels of nutrients, their absorption into the body will be poor if sufficient amounts of fat are not eaten along with the vegetables. The combination of a poor diet that is low in vegetables and not eating vegetables with sufficient fat therefore increases the likelihood of having low levels of vitamin E and vitamin K in the body where they are needed to promote health. Studies in humans clearly show that dietary fat is important for the absorption of vitamin E and vitamin K. However, limited information is available to indicate how much fat is optimal and whether fat specifically from eggs can help promote absorption of these nutrients. By successfully completing this study, we expect to demonstrate the benefits of eggs, by way of their fats found in the yolk, to improve the absorption of vitamin E and vitamin K that are naturally present in spinach.

## 2. How many people will take part in this study?

Our goal is to recruit healthy 10 men and women between the ages of 18-65 years. To meet this goal, we plan to screen up to 20 individuals.

## 3. What will happen if I take part in this study?

## **Screening**

Before participating in this study, you will need to visit our study center located in 219 Campbell Hall (1787 Neil Ave) on the Ohio State University campus for an initial blood screening to make sure you have fasting blood chemistries (glucose, triglyceride, cholesterol, hematocrit, and hemoglobin) that are consistent with our study criteria. During this time, an experienced technician will measure your blood pressure and collect a small blood sample (2 teaspoons) from your arm. Within a week, we will have determined your blood results, which we will provide to you. If your blood results are consistent with our study criteria, you will be eligible to continue with the study procedures. If not, you will not be able to participate in our study.

#### **Study Overview**

For this study, everyone will complete 6 separate nutrient absorption trials that are separated by at least 1 week. For 3 days prior to each nutrient absorption trial and the first day of each trial, we will be providing all of your foods and beverages. You will eat the same foods for each of the 6 nutrient absorption trials. During each trial, which will be completed over the course of 72 hours, you will receive a test meal containing spinach alone or in combination with eggs or other foods. Each test meal will be assigned by chance, but you will complete all test meals throughout the course of your participation in this study. If you are interested in

IRB Approval date:


2020)

learning about the final results of the study, we would be happy to email you a copy of the published study findings.

If you participate in this study, you will be scheduled at your convenience to visit our study center a total of 12 times after the initial screening meeting for the first trial, which includes picking up meals, having your height and weight measured, eating a test meal, and then allowing us to collect blood immediately before eating the test meal and then again at 3, 4.5, 6, 7.5, 9, 12, 24, 36, 48, and 72 hours after eating each test meal. You do not need to remain at our study center during this entire time and are free to leave between each study visit. For the 3 days prior and the first day of the study, we ask that you avoid consuming foods/drinks other than the ones we give to you. The amount of food given will be tailored to your caloric needs so that you maintain the same weight throughout the study. The meals will be cooked and ready to eat; a microwave may be used to reheat food if desired.

Additionally, the menus will be customized to your personal calorie level needed for weight maintenance. It is recommended (but not required) that you eat all that is provided to you so you maintain the same weight throughout the study. It is important to our study that you consume only the foods that we provide and not substitute any other foods without first discussing with the study coordinator. We will also give you a form to record any accidental intake of additional foods/drinks.

We also ask that you do not exercise for more than 7 hours per week throughout the entire study. For each morning visit to our study center, you will need to be fasted for 10-12 hours (no food or drink except for water). Please refer to the picture below for a visual overview of the study.



IRB Protocol Number: 2019H0504
IRB Approval date:


2020)

This study consists of 6 trials that are each 72 hours in duration. For each trial, you will visit the study center once approximately 3 days prior to starting the trial to pick up your foods and beverages. You will then visit the study center 11 times over 72 hours so we can collect a blood sample: 7 times on the first day, 2 times on the second day, 1 time on the third day, and 1 time on the fourth day. During each of these 11 blood draws, we will be collecting approximately 1 tablespoon of blood for each of the first 7 blood draws. For the remaining 4 blood draws, we will be collecting 0.5 tablespoons of blood each time. This will be approximately 0.6 cups of blood in total during each nutrient absorption trial. On the first day, you will also eat a test meal containing spinach alone (Trial 1), spinach with 1, 2, or 3 whole hardboiled eggs (Trials 2-4), spinach alone followed 1 egg 3 hours later (Trial 5), or spinach with 1 egg plus an additional egg 3 hours later (Trial 6).

For each morning visit on day 1, day 2, day 3, and day 4, we ask that you fast overnight for 10 hours, which means eating no foods or beverages other than water. After day 4, you can resume your normal daily activities. After about a week, we would like you to return to the study center to complete Trial 2. After this trial and another period of a week, you will return for Trial 3. After Trial 3 and another rest period of a week, you will return for Trial 4. After Trial 4 and another period of one week, you will return for Trial 5, and then after another rest period of about a week, you will return to the study center for Trial 6.

The below describes the procedures that will occur during each Trial.

**Study Visit 1.** This visit occurs approximately 3 days prior to your scheduled 72 hour nutrient absorption trial. Please return to our study center to pick up an insulated cooler containing your foods and beverages for the entire 3 days prior to starting your scheduled trial. This visit will be brief, no blood samples will be collected, and will last less than 15 minutes.

Study Visit 2 (Day 1 of Trial). We ask that you do not consume any food or drink except water for 10-12 hours prior to your study visit. Prior to providing you the test meal, we will measure your height, weight, waist circumference and blood pressure. We will then collect a 16 mL blood sample (1 tablespoon) for your 0 hour blood collection. You will then be asked to eat the test meal within 10 minutes. From that point, we ask that you remain in close proximity to our study center so that you may return for blood collection at 3, 4.5, 6, 9, 7.5 and 12 hours after eating the test meal. For each of these 6 blood draws, we will collect a 16 mL blood sample (1 tablespoon). On this day, we will also provide you lunch and dinner because it is important for our study to control your food intake. Each of the 7 blood collections during this day are expected to take less than 20 minutes.

Study Visit 3 (Day 2 of Trial). You will return to the study center after an overnight fast for blood collection that corresponds to 24 hours after you ate the test meal. You may then leave the study center. You will need to return at a time that corresponds to 36 hours after eating the test meal, but you do not need to be fasted. Both of the blood collections will be 8 mL each (half a tablespoon) are expected to take less than 20 minutes each.

IRB Protocol Number: 2019H0504
IRB Approval date:

rai uale.


2020)

Study Visit 4 (Day 3 of Trial). You will return to the study center after an overnight fast for blood collection that corresponds to 48 hours after you ate the test meal (8 mL or half a tablespoon of blood will be collected). You may then leave the study center and do not need to return again on this day. This blood collection is expected to take less than 20 minutes.

*Study Visit 5 (Day 4 of Trial).* You will return to the study center after an overnight fast for blood collection that corresponds to 72 hours after you ate the test meal (8 mL or half a tablespoon of blood will be collected). You may then leave the study center and do not need to return again on this day. This blood collection is expected to take less than 20 minutes.

#### **Blood Sample Storage Agreement**

Blood samples collected for this study will be analyzed for glucose, cholesterol, triglyceride, vitamin E, vitamin K, antioxidants (carotenoids and vitamin C), and measures related to inflammation (malondialdehyde). Any remaining samples, including those samples from individuals who do not meet eligibility requirements, will be stored up to 5 years at our study center. We ask that you allow us to store your samples for future analysis specifically related to this study. Storage of samples is completely optional and you may complete the study without agreeing to the storage of samples.

| , . | | s to store any remaining blood samples for a<br>sircle your response and provide your initials | |
|---|---|---|---|
| YES | NO | (Participant's Initials) | Date |
| 4 How k | ong will I b | o in the study? | |

# 4. How long will I be in the study?

You are required to visit the study center briefly at least 12 times per trial, for a total of 73 times to complete all 6 trials. Prior to joining the study, you will complete a screening visit, which will take about 1 hour. Visits in which you pick up food, eat test meals, and have blood collected are expected to take about 20 minutes each. Overall, we anticipate that you will commit about 21 hours over the course of about 12 weeks to complete the study, depending on your availability.

# 5. Can I stop being in the study?

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status. If you wish to have your samples destroyed, contact the investigator by phone or email.

IRB Protocol Number: IRB Approval date:


2020)

2019H0504

## 6. What risks, side effects or discomforts can I expect from being in the study?

The primary inconvenience for you is that you must visit our study center briefly 73 times over the course of the entire study. You will need to limit your exercise to less than 7 hours per week throughout the study. Additionally, you may consume only the food and beverage products provided to you for the 3 days prior and during the initial day of the study.

Blood Collection. During the blood drawing aspect of this investigation, only experienced technicians will be responsible for inserting all catheters and needles as well as collecting blood samples. All blood drawing materials will be sterile and sanitary techniques will be used. You may experience a small initial pain from insertion of the needle and bruising may occasionally occur after the procedures are completed. In addition, you may experience lightheadedness or feel faint which is common when people donate blood. During each trial, we will be collecting a total volume of 144 ml (~0.6 cup). Thus, 872 ml (~3.6 cups) of blood will be collected during the entire study (screening + 6 trials) that spans a minimum of 12 weeks. We advise participants not to donate blood and inform their doctor about the study if they need a blood draw at the doctor's office while they are on the study. We do not foresee any additional significant risks with collecting this amount of blood, other than the possible risks stated previously.

Spinach Test Meals. The test meals consist of spinach combined with hardboiled eggs. The spinach for this study will be grown special for this study using water that contains deuterium. Deuterium is a special type of hydrogen that is naturally found in water. It is being used because it is heavier than hydrogen typically found in water. This will allow the spinach to grow and produce vitamin E and vitamin K that contain deuterium. These forms of vitamin E and vitamin K can be measured in your blood after eating the spinach. With our laboratory instruments, we will be able to tell the difference between vitamin E and vitamin K from spinach versus all of the other foods that contain vitamin E and vitamin K from your diet. This allows us to measure absorption of these vitamins with high accuracy. The eggs used in these will be purchased form a local supermarket. There is no risk of eating cooked eggs, no additional risk of eating spinach that is grown with deuterium compared with spinach bought at the store, and no adverse effects are expected.

<u>Confidentiality.</u> To maintain your confidentiality, a number (i.e. code) will be assigned to you. This "code" will only be available to research personnel and any records containing your name will be stored in a locked filing cabinet within a lockable office or on a password protected computer in the principal investigator's laboratory or office. Research personnel under the supervision of the principal investigator and the principal investigator will be the only individuals that have access to this information.

## 7. What benefits can I expect from being in the study?

Although consumption of eggs with spinach is expected to have a positive effect, there is no guarantee the results will directly benefit you. You will be provided with your screening blood testing results as categorical information, because the results are for research purposes

Page 6 of 11

Form date: 05/17/2019

IRB Approval date:


2020)

and cannot be used to provide a clinical diagnosis of disease. In addition, we will provide information regarding your blood pressure, height, weight, waist circumference, and body mass index. If you are interested in learning more about your results during the study, we would be happy to email you a copy of the final study findings that are compiled in an anonymous manner once we have published our findings. Overall, the results obtained from this study are expected to enhance our knowledge of fat from eggs helps to improve the absorption of vitamin E and vitamin K that are naturally found in spinach. This knowledge is of great importance to increase our understanding of the potential health benefits of dietary patterns that link low-fat vegetables with other fat-containing foods to achieve appropriate levels of vitamins in our body.

## 8. What other choices do I have if I do not take part in the study?

You may choose not to participate without penalty or loss of benefits to which you are otherwise entitled.

## 9. Will my study-related information be kept confidential?

Efforts will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding study participation may be disclosed if required by state law.

Also, your records may be reviewed by the following groups (as applicable to the research):

- Office for Human Research Protections or other federal, state, or international regulatory agencies;
- U.S. Food and Drug Administration;
- The Ohio State University Institutional Review Board or Office of Responsible Research Practices;
- The sponsor supporting the study, their agents or study monitors; and
- Your insurance company (if charges are billed to insurance).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search the website at any time.

# 10. Will my de-identified information and bio-specimens be used or shared for future research?

Yes, they may be used or shared with other researchers without your additional informed consent.

IRB Approval date:


2020)

## 11. What are the costs of taking part in this study?

There will be no costs for participating in this study except those needed for transportation to and from the OSU campus.

## 12. Will I be paid for taking part in this study?

By law, payments to participants are considered taxable income. If you complete the study in its entirety and provide all requested blood samples and food-related records, and complete the four 72-hour nutrient absorption trials, you may receive up to \$450 (as a check) at the completion of the study. The check will be given at your final study visit. Parking for each visit following acceptance into the study will be paid for by a parking pass. For each of the trials following the informed consent and screening meeting, you will be paid in the following manner:

Trial 1 (Up to a total of \$12):

- \$1 will be provided for each of the 11 blood collections taking place over 72 hours (\$11 total)
- \$1 will be provided for food-related records (returning uneaten foods and/or empty containers)

Trial 2 (Up to a total of \$23):

- \$2 will be provided for each of the 11 blood collections taking place over 72 hours (\$22 total)
- \$1 will be provided for food-related records (returning uneaten foods and/or empty containers)

Trial 3 (Up to a total of \$45):

- \$4 will be provided for each of the 11 blood collections taking place over 72 hours (\$44 total)
- \$1 will be provided for food-related records (returning uneaten foods and/or empty containers)

Trial 4 (Up to a total of \$68):

- \$6 will be provided for each of the 11 blood collections taking place over 72 hours (\$66 total)
- \$2 will be provided for food-related records (returning uneaten foods and/or empty containers)

Trial 5 (Up to a total of \$90):

IRB Approval date:


2020)

• \$8 will be provided for each of the 11 blood collections taking place over 72 hours (\$88 total)

• \$2 will be provided for food-related records (returning uneaten foods and/or empty containers)

Trial 6 (Up to a total of \$112):

- \$10 will be provided for each of the 11 blood collections taking place over 72 hours (\$110 total)
- \$2 will be provided for food-related records (returning uneaten foods and/or empty containers)

#### Study Bonus:

If you complete the entire study and provide all of the requested materials, you will be provided \$350 plus a \$100 bonus, which will bring your total compensation to \$450. This will be given to you in the form of a check. If you withdraw or are dismissed from our study, you will be compensated for the completed aspects as indicated above.

## 13. What happens if I am injured because I took part in this study?

If you suffer an injury from participating in this study, you should notify the researcher or study doctor immediately, who will determine if you should obtain medical treatment at The Ohio State University Wexner Medical Center.

The cost for this treatment will be billed to you or your medical or hospital insurance. The Ohio State University has no funds set aside for the payment of health care expenses for this study.

IRB Approval date:


2020)

## 14. What are my rights if I take part in this study?

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights you may have as a participant in this study.

You will be provided with any new information that develops during the course of the research that may affect your decision whether or not to continue participation in the study.

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled.

An Institutional Review Board responsible for human subjects research at The Ohio State University reviewed this research project and found it to be acceptable, according to applicable state and federal regulations and University policies designed to protect the rights and welfare of research participants.

## 15. Who can answer my questions about the study?

For questions, concerns, or complaints about the study you may contact Dr. Richard Bruno (Principal Investigator; 614.292.5522; <a href="mailto:bruno.27@osu.edu">bruno.27@osu.edu</a>).

For questions about your rights as a participant in this study or to discuss other study-related concerns or complaints with someone who is not part of the research team, you may contact the Office of Responsible Research Practices at 1-800-678-6251.

If you are injured as a result of participating in this study or for questions about a study-related injury, you may contact Dr. Richard Bruno (Principal Investigator; 614.292.5522; bruno.27@osu.edu).

IRB Approval date:

Version: Ver 2 (Dec 7, 2020)

# Signing the consent form

I have read (or someone has read to me) this form and I am aware that I am being asked to participate in a research study. I have had the opportunity to ask questions and have had them answered to my satisfaction. I voluntarily agree to participate in this study.

I am not giving up any legal rights by signing this form. I will be given a copy of this form.

| Printed name of participant | Signature of participant |
|---|---|
| | AM/PM |
| | Date and time |
| Printed name of person authorized to consent for participant (when applicable) | Signature of person authorized to consent for participant (when applicable) |
| | AM/PM |
| Relationship to the participant | Date and time |
| A (D | |
| estigator/Research Staff | |
| ve explained the research to the participar | nt or his/her representative before requesting the |
| 1 1 | |
| nature(s) above. There are no blanks in thi | |
| | is document. A copy of this form has been given |
| · / | |
| · / | |
| ne participant or his/her representative. | is document. A copy of this form has been given |
| ne participant or his/her representative. | Signature of person obtaining consent AM/PM |
| ne participant or his/her representative. | Signature of person obtaining consent |
| Printed name of person obtaining consent | Signature of person obtaining consent Date and time AM/PM |
| ne participant or his/her representative. | Signature of person obtaining consent Date and time AM/PM |
| Printed name of person obtaining consent Witness(es) - May be left blank if not req | Signature of person obtaining consent Date and time Puired by the IRB |
| Printed name of person obtaining consent | Signature of person obtaining consent Date and time AM/PM |
| Printed name of person obtaining consent Witness(es) - May be left blank if not req | Signature of person obtaining consent Date and time Muired by the IRB Signature of witness AM/PM |
| Printed name of person obtaining consent Witness(es) - May be left blank if not req | Signature of person obtaining consent Date and time Date and time Signature of witness |
| Printed name of person obtaining consent Witness(es) - May be left blank if not req | Signature of person obtaining consent Date and time Muired by the IRB Signature of witness AM/PM |
| Printed name of person obtaining consent Witness(es) - May be left blank if not req Printed name of witness | Signature of person obtaining consent Date and time Signature of witness AM/PM Date and time AM/PM Date and time AM/PM |

IRB Approval date:


2020)

# The Ohio State University Consent to Participate in Research

Study Title: Achieving Nutritional Adequacy Of Vitamins E and K With An

Egg/Plant-Based Food Pairing – Study 2

**Principal Investigator:** Richard S. Bruno

**Sponsor:** Egg Nutrition Center / American Egg Board

• This is a consent form for research participation. It contains important information about this study and what to expect if you decide to participate. Please consider the information carefully. Feel free to discuss the study with your friends and family and to ask questions before making your decision whether or not to participate.

- Your participation is voluntary. You may refuse to participate in this study. If you decide to take part in the study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your usual benefits. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.
- You may or may not benefit as a result of participating in this study. Also, as explained below, your participation may result in unintended or harmful effects for you that may be minor or may be serious depending on the nature of the research.
- You will be provided with any new information that develops during the study that may affect your decision whether or not to continue to participate. If you decide to participate, you will be asked to sign this form and will receive a copy of the form. You are being asked to consider participating in this study for the reasons explained below.

#### **Key Information About This Study**

The following is a short summary to help you decide whether or not to be a part of this study. More detailed information is listed later in this form.

The purpose of this research is to understand how the absorption of vitamin E and vitamin K found in vegetables like spinach can be improved when eaten along with other foods like eggs that contain fat. If you choose to participate in this study, your involvement would span approximately 8 weeks. During this period, there will be 4 nutrient absorption trials. Each trial would last 72 hours and a trained individual would be collecting blood samples periodically from your arm (11 in total). However, you will be free to come and go from our study center during each trial. The primary risk in this study relates to the small initial pain, bruising, or lightheadedness you may experience during blood collection. There are no costs to you to participate in this research and benefits to you include receiving some of your blood testing results like glucose along with your blood pressure and body mass measurements.

IRB Approval date:


2020)

## 1. Why is this study being done?

Vitamin E and vitamin K are two important nutrients for human health. However, the majority of Americans eat diets that are lacking in these nutrients. In addition, when we eat vegetables containing these high levels of nutrients, their absorption into the body will be poor if sufficient amounts of fat are not eaten along with the vegetables. The combination of a poor diet that is low in vegetables and not eating vegetables with sufficient fat therefore increases the likelihood of having low levels of vitamin E and vitamin K in the body where they are needed to promote health. Studies in humans clearly show that dietary fat is important for the absorption of vitamin E and vitamin K. However, limited information is available to indicate how much fat is optimal and whether fat specifically from eggs can help promote absorption of these nutrients. By successfully completing this study, we expect to demonstrate the benefits of eggs, by way of their fats found in the yolk, to improve the absorption of vitamin E and vitamin K that are naturally present in spinach.

## 2. How many people will take part in this study?

Our goal is to recruit healthy 10 men and women between the ages of 18-65 years. To meet this goal, we plan to screen up to 20 individuals.

## 3. What will happen if I take part in this study?

## **Screening**

Before participating in this study, you will need to visit our study center located in 219 Campbell Hall (1787 Neil Ave) on the Ohio State University campus for an initial blood screening to make sure you have fasting blood chemistries (glucose, triglyceride, cholesterol, hematocrit, and hemoglobin) that are consistent with our study criteria. During this time, an experienced technician will measure your blood pressure and collect a small blood sample (2 teaspoons) from your arm. Within a week, we will have determined your blood results, which we will provide to you. If your blood results are consistent with our study criteria, you will be eligible to continue with the study procedures. If not, you will not be able to participate in our study.

#### **Study Overview**

For this study, everyone will complete 4 separate nutrient absorption trials that are separated by at least 1 week. For 3 days prior to each nutrient absorption trial and the first day of each trial, we will be providing all of your foods and beverages. You will eat the same foods for each of the 4 nutrient absorption trials. During each trial, which will be completed over the course of 72 hours, you will receive a test meal containing spinach in combination with eggs or other foods. Each test meal will be assigned by chance, but you will complete all test meals throughout the course of your participation in this study. If you are interested in

IRB Approval date:


2020)

learning about the final results of the study, we would be happy to email you a copy of the published study findings.

If you participate in this study, you will be scheduled at your convenience to visit our study center a total of 12 times after the initial screening meeting for the first trial, which includes picking up meals, having your height and weight measured, eating a test meal, and then allowing us to collect blood immediately before eating the test meal and then again at 3, 4.5, 6, 7.5, 9, 12, 24, 36, 48, and 72 hours after eating each test meal. You do not need to remain at our study center during this entire time and are free to leave between each study visit. For the 3 days prior and the first day of the study, we ask that you avoid consuming foods/drinks other than the ones we give to you. The amount of food given will be tailored to your caloric needs so that you maintain the same weight throughout the study. The meals will be cooked and ready to eat; a microwave may be used to reheat food if desired.

Additionally, the menus will be customized to your personal calorie level needed for weight maintenance. It is recommended (but not required) that you eat all that is provided to you so you maintain the same weight throughout the study. It is important to our study that you consume only the foods that we provide and not substitute any other foods without first discussing with the study coordinator. We will also give you a form to record any accidental intake of additional foods/drinks.

We also ask that you do not exercise for more than 7 hours per week throughout the entire study. For each morning visit to our study center, you will need to be fasted for 10-12 hours (no food or drink except for water). Please refer to the picture below for a visual overview of the study.

#### RANDOMIZATION SCHEME (N = 10 HEALTHY PERSONS)



Test meals will be assigned in random order, but each participant will complete 4 separate trials

#### For Each 72-Hour Nutrient Absorption Trial:

- ☐ Day 1: Eat assigned test meal and blood collected at 0, 3, 4.5, 6, 7.5, 9, 12 hours after the test meal
- ☐ Day 2: Blood collected at 24 hours and 36 hours after the test meal from Day 1
- □ Day 3: Blood collected at 48 hours after the test meal from Day 1
- □ Day 4: Blood collected at 72 hours after the test meal from Day 1

IRB Approval date:


2020)

This study consists of 4 trials that are each 72 hours in duration. For each trial, you will visit the study center once approximately 3 days prior to starting the trial to pick up your foods and beverages. You will then visit the study center 11 times over 72 hours so we can collect a blood sample: 7 times on the first day, 2 times on the second day, 1 time on the third day, and 1 time on the fourth day. During each of these 11 blood draws, we will be collecting approximately 1 tablespoon of blood at first 7 blood draws and 0.5 tablespoon of blood at rest 4 blood collections; or approximately 0.6 cups of blood in total during each nutrient absorption trial. On the first day, you will also eat a test meal containing spinach alone or in combination with whole hardboiled eggs, hardboiled egg whites, or vegetable oil. For each morning visit on day 1, day 2, day 3, and day 4, we ask that you fast overnight for 10 hours, which means eating no foods or beverages other than water. After day 4, you can resume your normal daily activities. After about a week, we would like you to return to the study center to complete Trial 2. After this trial and another period of a week, you will return for Trial 3 and then after another rest period of about a week, you will return to the study center for Trial 4.

The below describes the procedures that will occur during each Trial.

**Study Visit 1.** This visit occurs approximately 3 days prior to your scheduled 72 hour nutrient absorption trial. Please return to our study center to pick up an insulated cooler containing your foods and beverages for the entire 3 days prior to starting your scheduled trial. This visit will be brief, no blood samples will be collected, and will last less than 15 minutes.

Study Visit 2 (Day 1 of Trial). We ask that you do not consume any food or drink except water for 10-12 hours prior to your study visit. Prior to providing you the test meal, we will measure your height, weight, waist circumference and blood pressure. We will then collect a 16 mL blood sample (1 tablespoon) for your 0 hour blood collection. You will then be asked to eat the test meal within 10 minutes. From that point, we ask that you remain in close proximity to our study center so that you may return for blood collection at 3, 4.5, 6, 7.5, 9, and 12 hours after eating the test meal. For each of these 6 blood draws, we will collect a 16 mL blood sample (1 tablespoon). On this day, we will also provide you lunch and dinner because it is important for our study to control your food intake. Each of the 7 blood collections during this day are expected to take less than 20 minutes.

Study Visit 3 (Day 2 of Trial). You will return to the study center after an overnight fast for blood collection that corresponds to 24 hours after you ate the test meal. You may then leave the study center. You will need to return at a time that corresponds to 36 hours after eating the test meal, but you do not need to be fasted. Both of the blood collections will be 8 mL each (half a tablespoon) are expected to take less than 20 minutes each.

Study Visit 4 (Day 3 of Trial). You will return to the study center after an overnight fast for blood collection that corresponds to 48 hours after you ate the test meal (8 mL or half a tablespoon of blood will be collected). You may then leave the study center and do not need to return again on this day. This blood collection is expected to take less than 20 minutes.

CONSENT Biomedical/Cancer IRB Protocol Number: 2019H0504 IRB Approval date:


2020)

Study Visit 5 (Day 4 of Trial). You will return to the study center after an overnight fast for blood collection that corresponds to 72 hours after you ate the test meal (8 mL or half a tablespoon of blood will be collected). You may then leave the study center and do not need to return again on this day. This blood collection is expected to take less than 20 minutes.

#### **Blood Sample Storage Agreement**

Blood samples collected for this study will be analyzed for glucose, cholesterol, triglyceride, vitamin E, vitamin K, antioxidants (carotenoids and vitamin C), and measures related to inflammation (malondialdehyde). Any remaining samples, including those samples from individuals who do not meet eligibility requirements, will be stored up to 5 years at our study center. We ask that you allow us to store your samples for future analysis specifically related to this study. Storage of samples is completely optional and you may complete the study without agreeing to the storage of samples.

| , . | • | remaining blood samples for sponse and provide your initial | |
|---|---|---|---|
| YES | NO | (Participant's Initials) | Date |
| 4 TT 1 | | | |

## 4. How long will I be in the study?

You are required to visit the study center briefly at least 12 times per trial, for a total of 49 times to complete all 4 trials. Prior to joining the study, you will complete a screening visit, which will take about 1 hour. Visits in which you pick up food, eat test meals, and have blood collected are expected to take about 20 minutes each. Overall, we anticipate that you will commit about 14 hours over the course of about 8 weeks to complete the study, depending on your availability.

# 5. Can I stop being in the study?

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status. If you wish to have your samples destroyed, contact the investigator by phone or email.

## 6. What risks, side effects or discomforts can I expect from being in the study?

The primary inconvenience for you is that you must visit our study center briefly 49 times over the course of the entire study. You will need to limit your exercise to less than 7 hours per week throughout the study. Additionally, you may consume only the food and beverage products provided to you for the 3 days prior and during the initial day of the study.

CONSENT Biomedical/Cancer IRB Protocol Number: 2019H0504
IRB Approval date:


2020)

Blood Collection. During the blood drawing aspect of this investigation, only experienced technicians will be responsible for inserting all catheters and needles as well as collecting blood samples. All blood drawing materials will be sterile and sanitary techniques will be used. You may experience a small initial pain from insertion of the needle and bruising may occasionally occur after the procedures are completed. In addition, you may experience lightheadedness or feel faint which is common when people donate blood. During each trial, we will be collecting a total volume of 144 ml (~0.6 cup). Thus, 584 ml (~2.4 cups) of blood will be collected during the entire study (screening + 4 trials) that spans a minimum of 8 weeks. We advise participants not to donate blood and inform their doctor about the study if they need a blood draw at the doctor's office while they are on the study. We do not foresee any additional significant risks with collecting this amount of blood, other than the possible risks stated previously.

Spinach Test Meals. The test meals consist of spinach combined with hardboiled eggs. The spinach for this study will be grown special for this study using water that contains deuterium. Deuterium is a special type of hydrogen that is naturally found in water. It is being used because it is heavier than hydrogen typically found in water. This will allow the spinach to grow and produce vitamin E and vitamin K that contain deuterium. These forms of vitamin E and vitamin K can be measured in your blood after eating the spinach. With our laboratory instruments, we will be able to tell the difference between vitamin E and vitamin K from spinach versus all of the other foods that contain vitamin E and vitamin K from your diet. This allows us to measure absorption of these vitamins with high accuracy. The eggs used in these will be purchased form a local supermarket. There is no risk of eating cooked eggs, no additional risk of eating spinach that is grown with deuterium compared with spinach bought at the store, and no adverse effects are expected.

Confidentiality. To maintain your confidentiality, a number (i.e. code) will be assigned to you. This "code" will only be available to research personnel and any records containing your name will be stored in a locked filing cabinet within a lockable office or on a password protected computer in the principal investigator's laboratory or office. Research personnel under the supervision of the principal investigator and the principal investigator will be the only individuals that have access to this information.

## 7. What benefits can I expect from being in the study?

Although consumption of eggs with spinach is expected to have a positive effect, there is no guarantee the results will directly benefit you. You will be provided with your screening blood testing results as categorical information, because the results are for research purposes and cannot be used to provide a clinical diagnosis of disease. In addition, we will provide information regarding your blood pressure, height, weight, waist circumference, and body mass index. If you are interested in learning more about your results during the study, we would be happy to email you a copy of the final study findings that are compiled in an anonymous manner once we have published our findings. Overall, the results obtained from this study are expected to enhance our knowledge of fat from eggs helps to improve the

IRB Approval date:


2020)

absorption of vitamin E and vitamin K that are naturally found in spinach. This knowledge is of great importance to increase our understanding of the potential health benefits of dietary patterns that link low-fat vegetables with other fat-containing foods to achieve appropriate levels of vitamins in our body.

## 8. What other choices do I have if I do not take part in the study?

You may choose not to participate without penalty or loss of benefits to which you are otherwise entitled.

## 9. Will my study-related information be kept confidential?

Efforts will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding study participation may be disclosed if required by state law.

Also, your records may be reviewed by the following groups (as applicable to the research):

- Office for Human Research Protections or other federal, state, or international regulatory agencies;
- U.S. Food and Drug Administration;
- The Ohio State University Institutional Review Board or Office of Responsible Research Practices;
- The sponsor supporting the study, their agents or study monitors; and
- Your insurance company (if charges are billed to insurance).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search the website at any time.

# 10. Will my de-identified information and bio-specimens be used or shared for future research?

Yes, they may be used or shared with other researchers without your additional informed consent.

# 11. What are the costs of taking part in this study?

There will be no costs for participating in this study except those needed for transportation to and from the OSU campus.

## 12. Will I be paid for taking part in this study?

IRB Approval date:


2020)

By law, payments to participants are considered taxable income. If you complete the study in its entirety and provide all requested blood samples and food-related records, and complete the four 72-hour nutrient absorption trials, you may receive up to \$250 (as a check) at the completion of the study. The check will be given at your final study visit. Parking for each visit following acceptance into the study will be paid for by a parking pass. For each of the trials following the informed consent and screening meeting, you will be paid in the following manner:

#### Trial 1 (Up to a total of \$12):

- \$1 will be provided for each of the 11 blood collections taking place over 72 hours (\$11 total)
- \$1 will be provided for food-related records (returning uneaten foods and/or empty containers)

#### Trial 2 (Up to a total of \$23):

- \$2 will be provided for each of the 11 blood collections taking place over 72 hours (\$22 total)
- \$1 will be provided for food-related records (returning uneaten foods and/or empty containers)

#### Trial 3 (Up to a total of \$46):

- \$4 will be provided for each of the 11 blood collections taking place over 72 hours (\$44 total)
- \$2 will be provided for food-related records (returning uneaten foods and/or empty containers)

## Trial 4 (Up to a total of \$69 for grand total of \$150):

- \$6 will be provided for each of the 9 blood collections taking place over 72 hours (\$66 total)
- \$3 will be provided for food-related records (returning uneaten foods and/or empty containers)

#### Study Bonus:

If you complete the entire study and provide all of the requested materials, you will be provided a \$100 bonus, which will bring your total compensation to \$250. This will be given to you in the form of a check. If you withdraw or are dismissed from our study, you will be compensated for the completed aspects as indicated above.

## 13. What happens if I am injured because I took part in this study?

IRB Approval date:


2020)

If you suffer an injury from participating in this study, you should notify the researcher or study doctor immediately, who will determine if you should obtain medical treatment at The Ohio State University Wexner Medical Center.

The cost for this treatment will be billed to you or your medical or hospital insurance. The Ohio State University has no funds set aside for the payment of health care expenses for this study.

## 14. What are my rights if I take part in this study?

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights you may have as a participant in this study.

You will be provided with any new information that develops during the course of the research that may affect your decision whether or not to continue participation in the study.

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled.

An Institutional Review Board responsible for human subjects research at The Ohio State University reviewed this research project and found it to be acceptable, according to applicable state and federal regulations and University policies designed to protect the rights and welfare of research participants.

## 15. Who can answer my questions about the study?

For questions, concerns, or complaints about the study you may contact Dr. Richard Bruno (Principal Investigator; 614.292.5522; <u>bruno.27@osu.edu</u>).

For questions about your rights as a participant in this study or to discuss other study-related concerns or complaints with someone who is not part of the research team, you may contact the Office of Responsible Research Practices at 1-800-678-6251.

If you are injured as a result of participating in this study or for questions about a study-related injury, you may contact Dr. Richard Bruno (Principal Investigator; 614.292.5522; bruno.27@osu.edu).

IRB Approval date:


2020)

# Signing the consent form

I have read (or someone has read to me) this form and I am aware that I am being asked to participate in a research study. I have had the opportunity to ask questions and have had them answered to my satisfaction. I voluntarily agree to participate in this study.

I am not giving up any legal rights by signing this form. I will be given a copy of this form.

| Printed name of participant | Signature of participant |
|---|---|
| | AM/PI |
| | Date and time |
| Printed name of person authorized to consent for | Signature of person authorized to consent for participant |
| participant (when applicable) | (when applicable) |
| Relationship to the participant | AM/PN Date and time |
| tigator/Research Staff | |
| ature(s) above. There are no blanks in this participant or his/her representative. | nt or his/her representative before requesting the is document. A copy of this form has been given |
| ture(s) above. There are no blanks in thi | |
| ture(s) above. There are no blanks in thit participant or his/her representative. | Signature of person obtaining consent AM/PI |
| ature(s) above. There are no blanks in this participant or his/her representative. | Signature of person obtaining consent Date and time Am/P! |
| ature(s) above. There are no blanks in this e participant or his/her representative. Printed name of person obtaining consent | Signature of person obtaining consent Date and time Am/P! |
| ature(s) above. There are no blanks in this e participant or his/her representative. Printed name of person obtaining consent Witness(es) - May be left blank if not requ | Signature of person obtaining consent Date and time Puired by the IRB |
| Ature(s) above. There are no blanks in this participant or his/her representative. Printed name of person obtaining consent Witness(es) - May be left blank if not required. | Signature of person obtaining consent Date and time Puired by the IRB Signature of witness |
| Ature(s) above. There are no blanks in this participant or his/her representative. Printed name of person obtaining consent Witness(es) - May be left blank if not requ | Signature of person obtaining consent Date and time Puired by the IRB Signature of witness AM/PR |
| ature(s) above. There are no blanks in this e participant or his/her representative. Printed name of person obtaining consent Witness(es) - May be left blank if not requirement. Printed name of witness | Signature of person obtaining consent Date and time Signature of witness AM/P! Date and time AM/P! Date and time |

IRB Protocol Number:

IRB Approval date:

Version: Ver 1 (Jul 28,

2022)

2019H0504

# The Ohio State University Consent to Participate in Research

Study Title: Achieving Nutritional Adequacy Of Vitamins E and K With An

Egg/Plant-Based Food Pairing – Study 3

**Principal Investigator:** Richard S. Bruno

**Sponsor:** Egg Nutrition Center / American Egg Board

3

5

6

7

8

9

10

11

12

13

14

15

16

17 18

19

20

1 2

- This is a consent form for research participation. It contains important information about this study and what to expect if you decide to participate. Please consider the information carefully. Feel free to discuss the study with your friends and family and to ask questions before making your decision whether or not to participate.
- Your participation is voluntary. You may refuse to participate in this study. If you decide to take part in the study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your usual benefits. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.
- You may or may not benefit as a result of participating in this study. Also, as explained below, your participation may result in unintended or harmful effects for you that may be minor or may be serious depending on the nature of the research.
- You will be provided with any new information that develops during the study that may affect your decision whether or not to continue to participate. If you decide to participate, you will be asked to sign this form and will receive a copy of the form. You are being asked to consider participating in this study for the reasons explained below.

212223

24

#### **Key Information About This Study**

The following is a short summary to help you decide whether or not to be a part of this study. More detailed information is listed later in this form.

252627

28

29

30

31

32

3334

35

36

The purpose of this research is to understand how the absorption of vitamin E and vitamin K found in vegetables like spinach can be improved when eaten along with other foods like eggs that contain fat. If you choose to participate in this study, your involvement would span approximately 12 weeks. During this period, there will be 6 nutrient absorption trials. Each trial would last 72 hours and a trained individual would be collecting blood samples periodically from your arm (11 in total). However, you will be free to come and go from our study center during each trial. The primary risk in this study relates to the small initial pain, bruising, or lightheadedness you may experience during blood collection. There are no costs to you to participate in this research and benefits to you include receiving some of your blood testing results like glucose along with your blood pressure and body mass measurements.

IRB Protocol Number: IRB Approval date:

umber: 2019H0504 il date:

Version: Ver 1 (Jul 28, 2022)

## 1. Why is this study being done?

Vitamin E and vitamin K are two important nutrients for human health. However, the majority of Americans eat diets that are lacking in these nutrients. In addition, when we eat vegetables containing these high levels of nutrients, their absorption into the body will be poor if sufficient amounts of fat are not eaten along with the vegetables. The combination of a poor diet that is low in vegetables and not eating vegetables with sufficient fat therefore increases the likelihood of having low levels of vitamin E and vitamin K in the body where they are needed to promote health. Studies in humans clearly show that dietary fat is important for the absorption of vitamin E and vitamin K. However, limited information is available to indicate how much fat is optimal and whether fat specifically from eggs can help promote absorption of these nutrients. By successfully completing this study, we expect to demonstrate the benefits of eggs, by way of their fats found in the yolk, to improve the absorption of vitamin E and vitamin K that are naturally present in spinach.

## 2. How many people will take part in this study?

Our goal is to recruit up to 10 healthy men and women between the ages of 18-65 years. To meet this goal, we plan to screen up to 20 individuals.

## 3. What will happen if I take part in this study?

## Screening

Before participating in this study, you will need to visit our study center located in 219 Campbell Hall (1787 Neil Ave) on the Ohio State University campus for an initial blood screening to make sure you have fasting blood chemistries (glucose, triglyceride, cholesterol, hematocrit, and hemoglobin) that are consistent with our study criteria. During this time, an experienced technician will measure your blood pressure and collect a small blood sample (2 teaspoons) from your arm. Within a week, we will have determined your blood results, which we will provide to you. If your blood results are consistent with our study criteria, you will be eligible to continue with the study procedures. If not, you will not be able to participate in our

#### **Study Overview**

study.

For this study, everyone will complete 6 separate nutrient absorption trials that are separated by at least 1 week. For 3 days prior to each nutrient absorption trial and the first day of each trial, we will be providing all of your foods and beverages. You will eat the same foods for each of the 6 nutrient absorption trials. During each trial, which will be completed over the course of 72 hours, you will receive a test meal containing spinach alone or in combination with eggs or other foods. Each test meal will be assigned by chance, but you will complete all test meals throughout the course of your participation in this study. If you are interested in learning about

IRB Approval date:


2022)

the final results of the study, we would be happy to email you a copy of the published study findings.

80 81 82

83

84

85

86

87

88

89

90

79

If you participate in this study, you will be scheduled at your convenience to visit our study center a total of 12 times after the initial screening meeting for the first trial, which includes picking up meals, having your height and weight measured, eating a test meal, and then allowing us to collect blood immediately before eating the test meal and then again at 3, 4.5, 6, 7.5, 9, 12, 24, 36, 48, and 72 hours after eating each test meal. You do not need to remain at our study center during this entire time and are free to leave between each study visit. For the 3 days prior and the first day of the study, we ask that you avoid consuming foods/drinks other than the ones we give to you. The amount of food given will be tailored to your caloric needs so that you maintain the same weight throughout the study. The meals will be cooked and ready to eat; a microwave may be used to reheat food if desired.

91 92 93

94

95

96

97

Additionally, the menus will be customized to your personal calorie level needed for weight maintenance. It is recommended (but not required) that you eat all that is provided to you so you maintain the same weight throughout the study. It is important to our study that you consume only the foods that we provide and not substitute any other foods without first discussing with the study coordinator. We will also give you a form to record any accidental intake of additional foods/drinks.

98 99 100

101

102

We also ask that you do not exercise for more than 7 hours per week throughout the entire study. For each morning visit to our study center, you will need to be fasted for 10-12 hours (no food or drink except for water). Please refer to the picture below for a visual overview of the study.

103104

#### RANDOMIZATION SCHEME (N = 10 HEALTHY PERSONS) WASH-OUT WASH-OUT WASH-OUT TRIAL 1 TRIAL 2 TRIAL 3 TRIAL 4 ~1-WEEK ~1-WEEK ~1-WEEK Spinach O Eggs 1 Egg 2 Egg: WASH-OUT WASH-OUT ~1-WEEK TRIAL 5 TRIAL 6 ~1-WEEK Spinach Spinach 2 Egg whites Vegetable Oil

Test meals will be assigned in random order, but each participant will complete 6 separate trials

#### For Each 72-Hour Nutrient Absorption Trial:

- ☐ Day 1: Eat assigned test meal and blood collected at 0, 3, 4.5, 6, 7.5, 9, 12 hours after the test meal
- ☐ Day 2: Blood collected at 24 hours and 36 hours after the test meal from Day 1
- □ Day 3: Blood collected at 48 hours after the test meal from Day 1
- ☐ Day 4: Blood collected at 72 hours after the test meal from Day 1

IRB Protocol Number: IRB Approval date:

val date: Version: Ver 1 (Jul 28,

2022)

2019H0504

This study consists of 6 trials that are each 72 hours in duration. For each trial, you will visit the study center once approximately 3 days prior to starting the trial to pick up your foods and beverages. You will then visit the study center 11 times over 72 hours so we can collect a blood sample: 7 times on the first day, 2 times on the second day, 1 time on the third day, and 1 time on the fourth day. During each of these 11 blood draws, we will be collecting approximately 1 tablespoon of blood for each of the first 7 blood draws. For the remaining 4 blood draws, we will be collecting 0.5 tablespoons of blood each time. This will be approximately 0.6 cups of blood in total during each nutrient absorption trial. On the first day, you will also eat a test meal containing spinach alone (Trial 1), spinach with 1, 2, or 3 whole hardboiled eggs (Trials 2-4), spinach with two hardboiled egg whites (Trial 5), or spinach with vegetable oil (Trial 6).

For each morning visit on day 1, day 2, day 3, and day 4, we ask that you fast overnight for 10 hours, which means eating no foods or beverages other than water. After day 4, you can resume your normal daily activities. After about a week, we would like you to return to the study center to complete Trial 2. After this trial and another period of a week, you will return for Trial 3. After Trial 3 and another rest period of a week, you will return for Trial 4. After Trial 4 and another period of one week, you will return for Trial 5, and then after another rest period of about a week, you will return to the study center for Trial 6.

The below describes the procedures that will occur during each Trial.

**Study Visit 1.** This visit occurs approximately 3 days prior to your scheduled 72 hour nutrient absorption trial. Please return to our study center to pick up an insulated cooler containing your foods and beverages for the entire 3 days prior to starting your scheduled trial. This visit will be brief, no blood samples will be collected, and will last less than 15 minutes.

Study Visit 2 (Day 1 of Trial). We ask that you do not consume any food or drink except water for 10-12 hours prior to your study visit. Prior to providing you the test meal, we will measure your height, weight, waist circumference and blood pressure. We will then collect a 16 mL blood sample (1 tablespoon) for your 0 hour blood collection. You will then be asked to eat the test meal within 10 minutes. From that point, we ask that you remain in close proximity to our study center so that you may return for blood collection at 3, 4.5, 6, 7.5, 9, and 12 hours after eating the test meal. For each of these 6 blood draws, we will collect a 16 mL blood sample (1 tablespoon). On this day, we will also provide you lunch and dinner because it is important for our study to control your food intake. Each of the 7 blood collections during this day are expected to take less than 20 minutes.

Study Visit 3 (Day 2 of Trial). You will return to the study center after an overnight fast for blood collection that corresponds to 24 hours after you ate the test meal. You may then leave the study center. You will need to return at a time that corresponds to 36 hours after eating the test meal, but you do not need to be fasted. Both of the blood collections will be 8 mL each (half a tablespoon) are expected to take less than 20 minutes each.

CONSENT Biomedical/Cancer IRB Protocol Number: IRB Approval date:


2022)

2019H0504

Study Visit 4 (Day 3 of Trial). You will return to the study center after an overnight fast for blood collection that corresponds to 48 hours after you ate the test meal (8 mL or half a tablespoon of blood will be collected). You may then leave the study center and do not need to return again on this day. This blood collection is expected to take less than 20 minutes.

153154

155

156

**Study Visit 5 (Day 4 of Trial).** You will return to the study center after an overnight fast for blood collection that corresponds to 72 hours after you ate the test meal (8 mL or half a tablespoon of blood will be collected). You may then leave the study center and do not need to return again on this day. This blood collection is expected to take less than 20 minutes.

157158159

160

161

162

163

164

165

#### **Blood Sample Storage Agreement**

Blood samples collected for this study will be analyzed for glucose, cholesterol, triglyceride, vitamin E, vitamin K, antioxidants (carotenoids and vitamin C), and measures related to inflammation (malondialdehyde). Any remaining samples, including those samples from individuals who do not meet eligibility requirements, will be stored up to 5 years at our study center. We ask that you allow us to store your samples for future analysis specifically related to this study. Storage of samples is completely optional and you may complete the study without agreeing to the storage of samples.

166167168

169

Do you agree to allow us to store any remaining blood samples for additional future measurements? Please circle your response and provide your initials below:

170171172

YES NO

\_\_\_\_Date

173174

# 4. How long will I be in the study?

175176177

178

179

180

181

You are required to visit the study center briefly at least 12 times per trial, for a total of 73 times to complete all 6 trials. Prior to joining the study, you will complete a screening visit, which will take about 1 hour. Visits in which you pick up food, eat test meals, and have blood collected are expected to take about 20 minutes each. Overall, we anticipate that you will commit about 21 hours over the course of about 12 weeks to complete the study, depending on your availability.

(Participant's Initials)

182 183 184

# 5. Can I stop being in the study?

185 186

187

188

189

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status. If you wish to have your samples destroyed, contact the investigator by phone or email.

IRB Protocol Number:

IRB Approval date:


2022)

2019H0504

## 6. What risks, side effects or discomforts can I expect from being in the study?

192 193 194

195

196

198

199

200

201

202

203 204

205

206 207

208

The primary inconvenience for you is that you must visit our study center briefly 73 times over the course of the entire study. You will need to limit your exercise to less than 7 hours per week throughout the study. Additionally, you may consume only the food and beverage products

provided to you for the 3 days prior and during the initial day of the study. 197

Blood Collection. During the blood drawing aspect of this investigation, only experienced technicians will be responsible for inserting all catheters and needles as well as collecting blood samples. All blood drawing materials will be sterile and sanitary techniques will be used. You may experience a small initial pain from insertion of the needle and bruising may occasionally occur after the procedures are completed. In addition, you may experience lightheadedness or feel faint which is common when people donate blood. During each trial, we will be collecting a total volume of 144 ml (~0.6 cup). Thus, 872 ml (~3.6 cups) of blood will be collected during the entire study (screening + 6 trials) that spans a minimum of 12 weeks. We advise participants not to donate blood and inform their doctor about the study if they need a blood draw at the doctor's office while they are on the study. We do not foresee any additional significant risks with collecting this amount of blood, other than the possible risks stated previously.

Spinach Test Meals. The test meals consist of spinach combined with hardboiled eggs. The 209 spinach for this study will be grown special for this study using water that contains deuterium. 210 Deuterium is a special type of hydrogen that is naturally found in water. It is being used because 211 it is heavier than hydrogen typically found in water. This will allow the spinach to grow and 212 produce vitamin E and vitamin K that contain deuterium. These forms of vitamin E and vitamin 213 K can be measured in your blood after eating the spinach. With our laboratory instruments, we 214 will be able to tell the difference between vitamin E and vitamin K from spinach versus all of 215 the other foods that contain vitamin E and vitamin K from your diet. This allows us to measure 216 absorption of these vitamins with high accuracy. The eggs used in these will be purchased form 217 a local supermarket. There is no risk of eating cooked eggs, no additional risk of eating spinach 218 that is grown with deuterium compared with spinach bought at the store, and no adverse effects 219 are expected. 220

Confidentiality. To maintain your confidentiality, a number (i.e. code) will be assigned to you. This "code" will only be available to research personnel and any records containing your name will be stored in a locked filing cabinet within a lockable office or on a password protected computer in the principal investigator's laboratory or office. Research personnel under the supervision of the principal investigator and the principal investigator will be the only individuals that have access to this information.

227 228

221

222

223 224

225

226

# 7. What benefits can I expect from being in the study?

229 230

231

Although consumption of eggs with spinach is expected to have a positive effect, there is no guarantee the results will directly benefit you. You will be provided with your screening blood

IRB Protocol Number: IRB Approval date:

al date:

Version: Ver 1 (Jul 28, 2022)

2019H0504

testing results as categorical information, because the results are for research purposes and 232 cannot be used to provide a clinical diagnosis of disease. In addition, we will provide 233 information regarding your blood pressure, height, weight, waist circumference, and body mass 234 index. If you are interested in learning more about your results during the study, we would be 235 happy to email you a copy of the final study findings that are compiled in an anonymous manner 236 once we have published our findings. Overall, the results obtained from this study are expected 237 to enhance our knowledge of fat from eggs helps to improve the absorption of vitamin E and 238 vitamin K that are naturally found in spinach. This knowledge is of great importance to increase 239 our understanding of the potential health benefits of dietary patterns that link low-fat vegetables 240 with other fat-containing foods to achieve appropriate levels of vitamins in our body. 241

242243

## 8. What other choices do I have if I do not take part in the study?

244245

You may choose not to participate without penalty or loss of benefits to which you are otherwise entitled.

246247248

## 9. Will my study-related information be kept confidential?

249250

Efforts will be made to keep your study-related information confidential. However, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law.

252253254

251

Also, your records may be reviewed by the following groups (as applicable to the research):

255256

 Office for Human Research Protections or other federal, state, or international regulatory agencies;

257

• U.S. Food and Drug Administration;

258259

• The Ohio State University Institutional Review Board or Office of Responsible Research Practices;

260261

• Authorized Ohio State University staff not involved in the study may be aware that you are participating in a research study and have access to your information;

262263264

The sponsor supporting the study, their agents or study monitors; and
Your insurance company (if charges are billed to insurance).

266267

265

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search the website at any time.

268269

# 10. Will my de-identified information (and bio-specimens) be used or shared for future research?

270271272

Yes, it/they may be used or shared with other researchers without your additional informed consent.

IRB Protocol Number: 2019H0504 IRB Approval date:


2022)

## 11. What are the costs of taking part in this study?

275 276 277

There will be no costs for participating in this study except those needed for transportation to and from the OSU campus.

278 279 280

## 12. Will I be paid for taking part in this study?

281

282 By law, payments to participants are considered taxable income. If you complete the study in its entirety and provide all requested blood samples and food-related records, and complete the 283 four 72-hour nutrient absorption trials, you may receive up to \$450 (as a check) at the 284 completion of the study. The check will be given at your final study visit. Parking for each visit 285 following acceptance into the study will be paid for by a parking pass. For each of the trials 286 following the informed consent and screening meeting, you will be paid in the following 287

288 manner:

- Trial 1 (Up to a total of \$12): 289
- \$1 will be provided for each of the 11 blood collections taking place over 72 hours (\$11 290 total) 291
  - \$1 will be provided for food-related records (returning uneaten foods and/or empty containers)

293 294

292

- Trial 2 (Up to a total of \$23): 295
- \$2 will be provided for each of the 11 blood collections taking place over 72 hours (\$22 296 total)
- \$1 will be provided for food-related records (returning uneaten foods and/or empty 298 containers) 299

300

297

- Trial 3 (Up to a total of \$45): 301
- 302 \$4 will be provided for each of the 11 blood collections taking place over 72 hours (\$44 303
- \$1 will be provided for food-related records (returning uneaten foods and/or empty 304 containers) 305

306

- Trial 4 (Up to a total of \$68): 307
- \$6 will be provided for each of the 11 blood collections taking place over 72 hours (\$66 308 309 total)
- \$2 will be provided for food-related records (returning uneaten foods and/or empty 310 containers) 311

312

Trial 5 (Up to a total of \$90): 313

IRB Protocol Number: IRB Approval date:


2022)

2019H0504

• \$8 will be provided for each of the 11 blood collections taking place over 72 hours (\$88 total)

• \$2 will be provided for food-related records (returning uneaten foods and/or empty containers)

317318

316

- 319 Trial 6 (Up to a total of \$112):
- \$10 will be provided for each of the 11 blood collections taking place over 72 hours (\$110 total)
- \$2 will be provided for food-related records (returning uneaten foods and/or empty containers)

324

- 325 Study Bonus:
- If you complete the entire study and provide all of the requested materials, you will be provided \$350 plus a \$100 bonus, which will bring your total compensation to \$450. This will be given to you in the form of a check. If you withdraw or are dismissed from our study, you will be compensated for the completed aspects as indicated above.

329 330

13. What happens if I am injured because I took part in this study?

331332333

334

If you suffer an injury from participating in this study, you should notify the researcher or study doctor immediately, who will determine if you should obtain medical treatment at The Ohio State University Wexner Medical Center.

335336

The cost for this treatment will be billed to you or your medical or hospital insurance. The Ohio State University has no funds set aside for the payment of health care expenses for this study.

340341

14. What are my rights if I take part in this study?

342343

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights you may have as a participant in this study.

345346347

344

You will be provided with any new information that develops during the course of the research that may affect your decision whether or not to continue participation in the study.

348349

You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled.

- 353 An Institutional Review Board responsible for human subjects research at The Ohio State
- University reviewed this research project and found it to be acceptable, according to
- 355 applicable state and federal regulations and University policies designed to protect the rights
- and welfare of research participants.

CONSENT Biomedical/Cancer IRB Protocol Number: 2019H0504 IRB Approval date:


2022)

357 358

# 15. Who can answer my questions about the study?

359 360

For questions, concerns, or complaints about the study you may contact Dr. Richard Bruno (Principal Investigator; 614.292.5522; bruno.27@osu.edu).

361 362 363

364

For questions about your rights as a participant in this study or to discuss other study-related concerns or complaints with someone who is not part of the research team, you may contact the Office of Responsible Research Practices at 1-800-678-6251.

365 366 367

If you are injured as a result of participating in this study or for questions about a studyrelated injury, you may contact Dr. Richard Bruno (Principal Investigator; 614.292.5522; bruno.27@osu.edu).

369 370

| CONSENT |
|-------------------|
| Biomedical/Cancer |

IRB Protocol Number: 2019H0504
IRB Approval date:


2022)

| Signing the | consent | form |
|-------------|---------|------|
|-------------|---------|------|

372373

374

371

I have read (or someone has read to me) this form and I am aware that I am being asked to participate in a research study. I have had the opportunity to ask questions and have had them answered to my satisfaction. I voluntarily agree to participate in this study.

375376377

I am not giving up any legal rights by signing this form. I will be given a copy of this form.

| Printed name of participant | 6 |
|---|---|
| | Signature of participant |
| | AM/Pl |
| | Date and time |
| Printed name of person authorized to consent for participant (when applicable) | Signature of person authorized to consent for participant (when applicable) |
| · | |
| Relationship to the participant | Date and time AM/PI |
| Team on the participant | |
| Investigator/Research Staff | |
| in restiguest/iteseuren seum | |
| I have explained the research to the participan | t or his/her representative before requesting the |
| | s document. A copy of this form has been given |
| • • • • | s document. A copy of this form has been given |
| to the participant or his/her representative. | |
| Did I C III | - C: |
| Printed name of person obtaining consent | Signature of person obtaining consent |
| Printed name of person obtaining consent | |
| Printed name of person obtaining consent | |
| | Date and time |
| Printed name of person obtaining consent Witness(es) - May be left blank if not requ | Date and time |
| | Date and time |
| | Date and time |
| | Date and time |
| Witness(es) - May be left blank if not requ | Date and time tired by the IRB Signature of witness |
| Witness(es) - May be left blank if not requ | Date and time tired by the IRB Signature of witness AM/PN |
| Witness(es) - May be left blank if not requ | Date and time tired by the IRB Signature of witness |
| Witness(es) - May be left blank if not required name of witness | Date and time dired by the IRB Signature of witness AM/PM Date and time |
| Witness(es) - May be left blank if not requ | Date and time tired by the IRB Signature of witness Date and time Signature of witness |
| Witness(es) - May be left blank if not required name of witness | Date and time tired by the IRB Signature of witness AM/PN Date and time |